CLINICAL TRIAL: NCT03671356
Title: Risk Management in Interventional Cardiology - a Quality Management Single-center Registry
Acronym: NCDR
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 18-007
Record Dates: First submitted 2018-08-21; First posted 2018-09-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
Keywords: risk score; risk management; NCDR; interventional cardiology
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: risk score — risk score

SUMMARY:
The validity and applicability of different clinical risk scoring models in a variety of settings of interventional cardiology is evaluated in a retrospective and continuing prospective single-center registry at University Hospital Düsseldorf. Risk-adapted safety interventions are additionally tested.

DETAILED DESCRIPTION:
Beginning with a retrospective assessment of 2014-2017 and continuing with a prospective registry, clinical outcomes of interventional cardiac catheterization procedures at University Hospital Düsseldorf in a variety of settings (elective and emergency coronary procedures, structural and rhythmologic cardiac interventions etc.), will be evaluated. Different risk scoring models are recommended for risk stratification by cardiovascular societies (e.g. GRACE, CRUSADE, NCDR, ACEF, EUROScore scores) and will be evaluated for their applicability to contemporary and local clinical practice in interventional cardiology. Risk-adapted safety interventions (e.g. intensified monitoring, vascular access closure, renal protective measures) will be applied to all patients and will be evaluated for their impact on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >18 yeas of age, written informed consent, cardiac catheterization at university hospital Düsseldorf, Germany

Exclusion Criteria:

* no written informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consenting adult patients undergoing cardiac catheterization at University Hospital Düsseldorf, Germany
Sampling Method: Non-Probability Sample
Enrollment: 2067 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
mortality | 30 days
  In-hospital mortality will be assessed and primarily reported

SECONDARY OUTCOMES:
Bleeding (according to BARC bleeding definition) | 30 days and up to 5 years post procedure
  in-hospital and long-term minor and major bleeding up to five years post procedure will be assessed and reported
Acute and chronic kidney injury (according to KDIGO definitions) | 30 days and up to 5 years post procedure
  in-hospital and long-term acute and chronic kidney injury up to five years post procedure will be assessed and reported
TIA and Stroke | 30 days and up to 5 years post procedure
  in-hospital and long-term cerebrovascular events (TIA and stroke) up to five years post procedure will be assessed and reported
Quality of life (assessed by standardized QoL surveys) | 30 days and up to 5 years post procedure
  in-hospital and long-term impact of interventional procedures on quality of life up to five years post procedure will be assessed and reported
Long-term mortality | up to 5 years post procedure
  long-term mortality up to five years post procedure will be assessed and report

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Study Chair — Heinrich-Heine University, Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany